CLINICAL TRIAL: NCT05438914
Title: Subscapularis Repair in Reverse Shoulder Arthroplasty: a Randomized, Controlled, Multicenter, Prospective Study
Brief Title: Subscapularis Repair in Reverse Shoulder Arthroplasty
Acronym: Subscap
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AIRR-00608-20
Record Dates: First submitted 2022-05-19; First posted 2022-06-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Rotator Cuff Tear Arthropathy
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Intervention Model Description: The patients will be randomly allocated in a 1:1 ratio, with block sizes of four and six using a randomization sequence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Reverse Shoulder Arthroplasty with subscapularis repair (Experimental): The subscapularis will be repaired using the "suture through bone and prosthesis holes" surgical technique.
  Interventions: Device: Repair of the subscapularis
- Reverse Shoulder Arthroplasty without subscapularis repair (No Intervention): The subscapularis will not be repaired.

INTERVENTIONS:
Device: Repair of the subscapularis — The subscapularis will be repaired using the "suture through bone and prosthesis holes" surgical technique.
  Arms: Reverse Shoulder Arthroplasty with subscapularis repair

SUMMARY:
This study will evaluate the subscapularis repair versus non-repair during a reverse shoulder arthroplasty (RSA).

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate pain and function in patients undergoing RSA with or without subscapularis repair. This primary outcome will be measured by analysis of Constant scores at two years post-operative.

Secondary objectives are to evaluate pain, function and imaging, between the two groups at each applicable time point.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is scheduled to undergo a reverse shoulder arthroplasty procedure using the Arthrex ReversTM system.
2. Patient voluntarily consents to participate in the study and has the mental and physical ability to participate in the study, fill out subjective questionnaires, return for follow-up visits, and comply with prescribed post-operative physical therapy.
3. Patient meets FDA cleared indications for reverse shoulder arthroplasty
4. Patient is between 18-100 years old
5. Patient agrees to also be enrolled in the Arthrex Total Shoulder Registry Study
6. Patient has a standard of care pre-operative CT taken within 6 months that has been submitted for Arthrex Virtual Implant Positioning TM (VIP) planning

Exclusion Criteria:

1. Patient has a history of ipsilateral shoulder arthroplasty
2. A history of shoulder septic arthritis
3. A full thickness subscapularis tear
4. An acute or malunited proximal humeral fracture
5. Chronic locked dislocation
6. Rheumatoid arthritis
7. Tumors
8. Axillary nerve damage
9. Non-functioning deltoid muscle
10. Glenoid vault deficiency precluding baseplate fixation
11. Infection and neuropathic joints
12. Known or suspected non-compliance, drug or alcohol abuse
13. Patients incapable of judgement or under tutelage
14. Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, contraindication for imaging etc.
15. The subject is related to investigator as family members, employees, or other dependent persons
16. Any prior open anterior shoulder surgery that included takedown of the subscapularis tendon or violation of the subscapularis tendon (i.e. Latarjet, Bristow)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2025-09-14 (Estimated); Study Completion 2025-09-14 (Estimated)

PRIMARY OUTCOMES:
Constant-Murley Shoulder Outcome Score | Collected at at pre-op, but the primary outcome is the score at 2 years post-procedure.
  A combination of objective measures and patient-reported outcomes. It defines the level of pain and the ability to carry out the normal daily activities of the patient. It is a 0-100 point scale, the higher the score, the higher the quality of the function.
Constant-Murley Shoulder Outcome Score | Collected at at 9 week post-op timepoint, but the primary outcome is the score at 2 years post-procedure.
  A combination of objective measures and patient-reported outcomes. It defines the level of pain and the ability to carry out the normal daily activities of the patient. It is a 0-100 point scale, the higher the score, the higher the quality of the function.
Constant-Murley Shoulder Outcome Score | Collected at at the 26 week post-op timepoint, but the primary outcome is the score at 2 years post-procedure.
  A combination of objective measures and patient-reported outcomes. It defines the level of pain and the ability to carry out the normal daily activities of the patient. It is a 0-100 point scale, the higher the score, the higher the quality of the function.
Constant-Murley Shoulder Outcome Score | Collected at at 1 year post-op timepoint, but the primary outcome is the score at 2 years post-procedure.
  A combination of objective measures and patient-reported outcomes. It defines the level of pain and the ability to carry out the normal daily activities of the patient. It is a 0-100 point scale, the higher the score, the higher the quality of the function.
Constant-Murley Shoulder Outcome Score | Collected at the 2 year post-op timepoint, and is the primary outcome measure
  A combination of objective measures and patient-reported outcomes. It defines the level of pain and the ability to carry out the normal daily activities of the patient. It is a 0-100 point scale, the higher the score, the higher the quality of the function.

SECONDARY OUTCOMES:
Ultrasound | Collected once at either the 6 month, 1 year or 2 year timepoint.
  Evaluation of the subscapularis complex in patients that have been randomized to "repair of the subscapularis" to examine the subscapularis complex. Ultrasound scans will be read and the integrity of the subscapularis complex will be determined by the clinician to be "intact", "attenuated", "partial tear" or "complete tear".
American Shoulder and Elbow Surgeons (ASES) subjective survey | Collected at pre-op, 9 weeks, 26 weeks, 1 year and 2 year post-op timepoints.
  A combination of objective measures and patient-reported outcomes, it measures pain and functional limitations in the shoulder. The objective questionnaire allows documentation of range of motion in the patient.
Simple Shoulder Test (SST) questionnaire | Collected at pre-op, 9 weeks, 26 weeks, 1 year and 2 year post-op timepoints.
  Provides a standardized way of recording the function of a shoulder before and after treatment.
Visual Analog Scale (VAS) | Collected at pre-op, 9 weeks, 26 weeks, 1 year and 2 year post-op timepoints.
  The standard measure for pain on a 0-10 scale, 10 being the worst.
Western Ontario Osteoarthritis of the Shoulder Index (WOOS) | Collected at pre-op, 9 weeks, 26 weeks, 1 year and 2 year post-op timepoints.
  A patient administrated questionnaire for measurement of the quality of life. It provides scores on four domains: 1.) physical symptoms, 2.) sport, recreation, and work, 3.) lifestyle and 4.) emotions.
Veterans Rand 12 Item Health Survey (VR-12) | Collected at pre-op, 9 weeks, 26 weeks, 1 year and 2 year post-op timepoints.
  A self-administered health measure. Answers are summarized into two scores, a Physical Component Score and a Mental Component Score, which provides an important contrast between the respondents' physical and psychological health status.
Single Assessment Numeric Evaluation score (SANE) | Collected at pre-op, 9 weeks, 26 weeks, 1 year and 2 year post-op timepoints.
  Asks patients to rate shoulder pain as a percentage of normal.
Standard Pre-Operative Form | Collected at the pre-op visit.
  A patient administered form that asks patients to evaluate their expectations of their scheduled Arthroplasty procedure.
Return to Work Form | Collected at pre-op, 26 weeks and 1 year.
  A patient administered form that asks patients to determine the effect that their shoulder has had on their employment.
Standard Late Postoperative Form | Collected at the 1 year and 2 year timepoints.
  A patient administered form that asks patient to evaluate if their expectations were met regarding their Arthroplasty procedure.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - The University of Arizona/Banner Health, Phoenix, Arizona
  - Western Orthopaedics, P.C., Denver, Colorado
  - Southern Oregon Orthopedics, Medford, Oregon
  - The Hawkins Foundation, Greenville, South Carolina
  - The Campbell Clinic, Collierville, Tennessee
  - Jordan Young Institute, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No